CLINICAL TRIAL: NCT02982707
Title: Single-dose Pharmacokinetics of BMS-986177 in Participants With Hepatic Impairment Compared to Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV010-013
Record Dates: First submitted 2016-11-15; First posted 2016-12-05 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — milvexian

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mild Hepatic Subjects (Experimental): Subjects are given a single dose of BMS-986177
  Interventions: Drug: BMS-986177
- Moderate Hepatic Subjects (Experimental): Subjects are given a single dose of BMS-986177
  Interventions: Drug: BMS-986177
- Healthy Match Subjects (Experimental): Subjects are given a single dose of BMS-986177
  Interventions: Drug: BMS-986177

INTERVENTIONS:
Drug: BMS-986177 — Single oral dose

SUMMARY:
A single oral dose of BMS-986177 administered to subjects of mild hepatic impairment, moderate hepatic impairment and healthy matched subjects to evaluate pharmacokinetics, safety, and tolerability in these subjects

ELIGIBILITY:
Inclusion Criteria:

* Women not of childbearing potential (WNOCBP) and males. Women must have documented proof they are not of childbearing potential
* BMI of 20.0 to 38.0 kg/m2, inclusive
* Hepatic subjects classified as Child-Pugh mild (Class A) or Child-Pugh moderate (Class B) who have had no significant change to disease status in past 6 months and are on stable treatment regimen
* Healthy subjects must not have clinically significant deviations from normal in medical history, physical exam, ECGs, vital signs or clinical lab values

Exclusion Criteria:

* Evidence of coagulopathy, prolonged or unexplained clinically significant bleeding, or frequent unexplained bruising or thrombus formation
* Use of corticosteroids, nonsteroidal anti-inflammatory compounds, aspirin or other antiplatelet agents or anticoagulants within 2 weeks of dosing
* Healthy subjects must not have used tobacco or have a history of drug or alcohol abuse within the last 6 months
* Subjects must not have a current or recent (within 3 months) GI disease that increases participant risk of GI bleeding or interferes with absorption of the study drug

Other protocol defined inclusion and exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986177 | Up to 5 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) of BMS-987177 | Up to 5 days
Area under the plasma concentration-time curve from time zero to the time the last quantifiable concentration (AUC(0-T)) of BMS-986177 | Up to 5 days
Area under the plasma concentration-time curve from time zero to (AUC(0-72)) of BMS-986177 | Up to 5 days

SECONDARY OUTCOMES:
Incidence of adverse events (AEs), serious adverse events (SAEs), and AEs leading to discontinuation | Screening until 30 days after discontinuation of dosing or subject's participation
Number of participants with clinical laboratory abnormalities | Screening until 30 days after discontinuation of dosing or subject's participation
Number of participants with clinically significant changes in electrical activity of the heart measured by electrocardiogram (ECG) | Screening until 30 days after discontinuation of dosing or subject's participation
Number of participants with vital sign abnormalities | Screening until 30 days after discontinuation of dosing or subject's participation

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Texas Liver Institute, San Antonio, Texas

REFERENCES:
- [Derived] Perera V, Abelian G, Li D, Wang Z, Zhang L, Lubin S, Chen W, Bello A, Murthy B. Single-Dose Pharmacokinetics of Milvexian in Participants with Mild or Moderate Hepatic Impairment Compared with Healthy Participants. Clin Pharmacokinet. 2022 Jun;61(6):857-867. doi: 10.1007/s40262-022-01110-9. Epub 2022 Mar 9. PMID 35262846
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Education Resource — https://www.bmsstudyconnect.com/s/US/English/USenHome